CLINICAL TRIAL: NCT07126652
Title: Serological Responses to Adjuvanted Versus Non-adjuvanted Influenza Vaccines Among People With HIV: a Randomized Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University Hospital, Cancer Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 202506103MIPD
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: Antibody Response
Keywords: HIV; influenza; vaccination; MF-59
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MF-59 (Experimental)
  Interventions: Drug: MF-59
- Cell-based (Active Comparator)
  Interventions: Drug: cell-based
- Egg-based (Active Comparator)
  Interventions: Drug: egg-based

INTERVENTIONS:
Drug: MF-59 — MF-59 influenza vaccination
  Arms: MF-59
Drug: cell-based — cell-based influenza vaccination
  Arms: Cell-based
Drug: egg-based — egg-based influenza vaccination
  Arms: Egg-based

SUMMARY:
Until now, the adjuvanted influenza-related studies focused mainly on people at older ages. However, the data on immunocompromised people, who might have suboptimal serological responses when receiving nonadjuvanted vaccines, is scarce. In this study, we aim to compare the immunogenicity and safety to adjuvanted versus nonadjuvanted seasonal influenza vaccines among people with HIV.

ELIGIBILITY:
Inclusion Criteria:

* People with HIV aged > 50 years
* Latest HIV RNA load tested less than 330 IU/mL

Exclusion Criteria:

* Confirmed serious adverse effect owing to any type of inluenza vaccine
* severe coagulopathy
* Have recieved influenza vaccine of 2025-2026 season

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
SCR | between Day 1 and Day 28±7.
  The primary end point includes SCR measured by the change in HI titer in serum against the vaccine strains between Day 1 and Day 28±7.

IPD SHARING:
Plan to Share IPD: No